CLINICAL TRIAL: NCT03351777
Title: Efficacy and Safety of PR022 Topical Gel to Treat Mild-to-Moderate Atopic Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Realm Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REALM-1
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PR022 topical gel, 0.05% (Experimental): Applied twice daily for 28 days
  Interventions: Drug: PR022
- PR022 topical gel, 0.1% (Experimental): Applied twice daily for 28 days
  Interventions: Drug: PR022
- PR022 topical gel vehicle (Placebo Comparator): Applied twice daily for 28 days
  Interventions: Drug: PR022

INTERVENTIONS:
Drug: PR022 — Topical Gel

SUMMARY:
The purpose of this study is to determine whether PR022 Topical Gels are safe and effective treatments for mild-to-moderate atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 to 65 years of age
* EASI score ≤ 21 at baseline
* Diagnosis of mild-to-moderate (grade 2 or 3) AD according to the ISGA scale at Baseline
* BSA affected by AD: 5% to 20% at start of treatment
* Willing and able to apply study treatments as directed, comply with study instructions, and commit to attending all visits
* Willing and able to provide informed consent
* Use of adequate birth control, if of reproductive potential and sexually active

Exclusion Criteria:

* Widespread AD requiring systemic therapy
* Use of any of the following treatments within the specified time periods prior to Day 1
* Topical medications (topical antibiotics, topical corticosteroids, topical antifungals, topical antihistamines, topical retinoids, topical calcipotriene, tacrolimus, pimecrolimus, or other topical drug products for treatment of AD) or bleach bath within 2 weeks prior to Day 1
* Systemic agents (cyclosporine, systemic corticosteroids [oral and injectable; intranasal and inhaled corticosteroids are allowed if use is kept constant during the study], systemic antibiotics, immunomodulators or immunosuppressive therapies, interferon, cytotoxic drugs [e.g., methotrexate, cyclophosphamide, azathioprine], oral retinoids, systemic antifungals, tacrolimus) for the treatment of AD within 4 weeks prior to Day 1
* Ultraviolet (UV) therapy or use of a tanning booth/parlor within 6 weeks prior to Day 1
* Biologic therapies within 12 weeks (or 5 half-lives) prior to Day 1
* Antihistamines within 5 days prior to Day 1 [stable regimens (consistent use ≥ 14 days before Day 1) of oral H1 antihistamines for non-AD lesion treatment will be allowed]
* Active or potentially recurrent dermatologic condition other than AD that may confound evaluation
* Congenital ichthyosis (note that subjects with ichthyosis vulgaris are permitted)
* Known allergy to any ingredients of the investigational product formulation
* Significant confounding conditions as assessed by Investigator
* Any condition that could interfere with any evaluation in the study
* Pregnancy or breast feeding
* Any reason which, in the opinion of the Investigator, interferes with the ability of the subject to participate in or complete the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Percent change from Baseline to Day 29 in Eczema Area and Severity Index (EASI) | 29 days

SECONDARY OUTCOMES:
Percentage of subjects who achieved success in Investigator's Static Global Assessment (ISGA), defined as a score of "Clear" (0) or "Almost Clear" (1) with a minimum 2-grade improvement at Day 29 | 29 Days
Percentage of subjects with an ISGA score of "Clear" (0) or "Almost Clear" (1) at Day 29 | 29 Days
Percentage of subjects with EASI-75 (≥ 75% improvement from Baseline) at Day 29 | 29 Days
Percentage of subjects with EASI-50 (≥ 50% improvement from Baseline) at Day 29 | 29 Days
Percent change from Baseline to Day 29 in body surface area (BSA) affected by AD | 29 Days
Change from Baseline to Day 29 in SCORing Atopic Dermatitis (SCORAD) | 29 Days
Percent change from Baseline to Day 29 in pruritus Numerical Rating Scale (NRS) | 29 Days
Change from Baseline to Day 29 in 5 dimensions of itch (5-D Itch) scale | 29 days
Change from Baseline to Day 29 in Dermatology Life Quality Index (DLQI) | 29 days
Frequency counts and percentages of DLQI scores (scored 0 to 3) at Baseline and Day 29, as well as shift in DLQI scores from Baseline to Day 29 | 29 Days

OTHER OUTCOMES:
Change in serum IgE titer and TARC concentration from Baseline to Day 29 | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Peters, MD, PhD, Study Director — Realm
Locations (1):
- Principal Investigator, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided